CLINICAL TRIAL: NCT04642716
Title: Evaluation of Free Aminoacids in Saliva as A Diagnostic Biomarker of Periodontal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Nur Balci, DDs, PhD, Dr. Nur Balci, Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10840098-327
Record Dates: First submitted 2020-11-20; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Periodontitis; Diagnoses Disease
Keywords: Saliva; Amino acids; Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Saliva of periodontitis patients collected for analyzing free amino acids.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Salivary free amino acids profile observation (Other): Saliva samples of periodontitis patients and healthy controls were collected. The AA analysis of the saliva was performed by LC-MS/MS by using the Thermo Scientific TSQ Quantum Access MAX (Thermo Scientific, Schaumburg, IL, USA) .
  Interventions: Other: Saliva collection of patients and salivary free amino acids analysis

INTERVENTIONS:
Other: Saliva collection of patients and salivary free amino acids analysis
  Other Names: Salivary free amino acids in patients with periodontitis

SUMMARY:
Amino acids (AAs) are organic molecules that are associated with inflammation and innate immunity diseases with critical roles in the cell repair and protection process. Our aim was to identify the free amino acids in saliva of a group of periodontitis patients and healthy individuals and additionally to assess their levels in different periodontal disease types and compare it to the healthy individuals.

DETAILED DESCRIPTION:
The study consisted of three groups: healthy individuals (control(C); n=20), Stage III Grade B generalized periodontitis (GP-B; n=20), and Stage III Grade C generalized periodontitis (GP-C; n=20). Clinical periodontal parameters (plaque index (PI), gingival index (GI), probing depth (PPD), gingival recession (GR), clinical attachment level (CAL) and bleeding on probing (BOP)) were measured. The amino acid analysis in saliva was accomplished by liquid chromatography-mass spectrometry (LC MS/MS) as mean concentration.

ELIGIBILITY:
Inclusion Criteria:

systemically healthy, clinical diagnosis of periodontitis, clinical diagnosis of periodontal health

Exclusion Criteria:

history of regular use of systemic antibiotics, anti-inflammatory, or antioxidant drugs (previous 3 months); nonsurgical periodontal treatment (previous 6 months); surgical periodontal treatment (previous 12 months); presence of <10 teeth; current medications affecting gingival health (calcium channel blockers, phenytoin, cyclosporine, and hormone replacement therapy); diabetes diagnosis; rheumatoid arthritis diagnosis; and pregnancy, lactating, smoking, or excessive alcohol consumption.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-08-03 (Actual)

PRIMARY OUTCOMES:
Pocket probing depth | 2 years
  Measurement of the depth of a sulcus or periodontal pocket determined by measuring distance from a gingival margin to the base of the sulcus or pocket with a calibrated periodontal probe.
Clinical attachment level | 2 years
  Clinical attachment level (or loss, CAL) is a more accurate indicator of the periodontal support around a tooth than probing depth alone. CAL is measured from a fixed point on the tooth that does not change, the CEJ.
  To calculate CAL, two measurements are needed: distance from the gingival margin to the CEJ and probing depth.
  In recession: probing depth (+) gingival margin to the CEJ (add). In tissue overgrowth: probing depth (-) gingival margin to the CEJ (subtract)
Bleeding on probing | 2 years
  referring to bleeding that is induced by gentle manipulation of the tissue at the depth of the gingival sulcus, or interface between the gingiva and a tooth.

SECONDARY OUTCOMES:
Amino acid Analysis | 2 years
  The AA analysis of the saliva was performed by LC-MS/MS by using the Thermo Scientific TSQ Quantum Access MAX (Thermo Scientific, Schaumburg, IL, USA) according to a modified version of Le et al.'s method.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erratum for Wang et al. Glycine stimulates protein synthesis and inhibits oxidative stress in pig small intestinal epithelial cells. J Nutr 2014;144:1540-8. J Nutr. 2016 Sep;146(9):1813. doi: 10.3945/jn.116.236612. No abstract available. PMID 27587752
- [Background] Li P, Yin YL, Li D, Kim SW, Wu G. Amino acids and immune function. Br J Nutr. 2007 Aug;98(2):237-52. doi: 10.1017/S000711450769936X. Epub 2007 Apr 3. PMID 17403271
- [Background] Cruzat VF, Krause M, Newsholme P. Amino acid supplementation and impact on immune function in the context of exercise. J Int Soc Sports Nutr. 2014 Dec 14;11(1):61. doi: 10.1186/s12970-014-0061-8. eCollection 2014. PMID 25530736
- [Background] Song Zh, Tong G, Xiao K, Jiao le F, Ke Yl, Hu Ch. L-cysteine protects intestinal integrity, attenuates intestinal inflammation and oxidant stress, and modulates NF-kappaB and Nrf2 pathways in weaned piglets after LPS challenge. Innate Immun. 2016 Apr;22(3):152-61. doi: 10.1177/1753425916632303. Epub 2016 Feb 25. PMID 26921254
- [Background] Sido B, Seel C, Hochlehnert A, Breitkreutz R, Droge W. Low intestinal glutamine level and low glutaminase activity in Crohn's disease: a rational for glutamine supplementation? Dig Dis Sci. 2006 Dec;51(12):2170-9. doi: 10.1007/s10620-006-9473-x. Epub 2006 Nov 1. PMID 17078002
- [Background] Onder C, Kurgan S, Altingoz SM, Bagis N, Uyanik M, Serdar MA, Kantarci A, Gunhan M. Impact of non-surgical periodontal therapy on saliva and serum levels of markers of oxidative stress. Clin Oral Investig. 2017 Jul;21(6):1961-1969. doi: 10.1007/s00784-016-1984-z. Epub 2016 Nov 2. PMID 27807715
- [Background] Dede FO, Ozden FO, Avci B. 8-hydroxy-deoxyguanosine levels in gingival crevicular fluid and saliva in patients with chronic periodontitis after initial periodontal treatment. J Periodontol. 2013 Jun;84(6):821-8. doi: 10.1902/jop.2012.120195. Epub 2012 Aug 16. PMID 22897655
- [Background] Rajda C, Tajti J, Komoroczy R, Seres E, Klivenyi P, Vecsei L. Amino acids in the saliva of patients with migraine. Headache. 1999 Oct;39(9):644-9. doi: 10.1046/j.1526-4610.1999.3909644.x. PMID 11279959
- [Background] Le A, Ng A, Kwan T, Cusmano-Ozog K, Cowan TM. A rapid, sensitive method for quantitative analysis of underivatized amino acids by liquid chromatography-tandem mass spectrometry (LC-MS/MS). J Chromatogr B Analyt Technol Biomed Life Sci. 2014 Jan 1;944:166-74. doi: 10.1016/j.jchromb.2013.11.017. Epub 2013 Nov 18. PMID 24316529
- [Derived] Balci N, Kurgan S, Cekici A, Cakir T, Serdar MA. Free amino acid composition of saliva in patients with healthy periodontium and periodontitis. Clin Oral Investig. 2021 Jun;25(6):4175-4183. doi: 10.1007/s00784-021-03977-7. Epub 2021 May 11. PMID 33977387